CLINICAL TRIAL: NCT05045599
Title: Effectiveness of Integrating Family Planning - Maternal, Newborn and Child Health (MNCH) Services on Uptake of Voluntary Modern Contraceptive Methods in Rural District of Sindh Province: A Quasi-experimental Study
Brief Title: Effectiveness of Integrating Family Planning - Maternal, Newborn and Child Health (MNCH) Services on Uptake of Voluntary Modern Contraceptive Methods
Acronym: RMNCH FP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aga Khan University (Other)
Collaborators: United Nations (Other); Global Affairs Canada (Other)
Responsible Party: Principal Investigator, Dr Zulfiqar Ahmed Bhutta, Distinguished University Professor, Aga Khan University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-3606-18261-1
Record Dates: First submitted 2021-09-07; First posted 2021-09-16 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Reproductive Behavior, Family Planning Services
Keywords: RMNCH, FP
MeSH Terms: conditions — Reproductive Behavior | interventions — Child Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Integration of Family planning in Maternal, Newborn and Child Health (Experimental): Strengthening of capacity of LHWs and Health care provider in providing integrated services Ensure Sustained supplies are available Community Mobilization Infrastructure support to ensure privacy and confidentiality Improvement of data recording, reporting and use
  Interventions: Behavioral: Capacity Building of Health care workers and providers to deliver integrated Family Planning and Maternal, Newborn and Child Health
- Standard of care (Active Comparator)
  Interventions: Behavioral: Capacity Building of Health care workers and providers to deliver integrated Family Planning and Maternal, Newborn and Child Health

INTERVENTIONS:
Behavioral: Capacity Building of Health care workers and providers to deliver integrated Family Planning and Maternal, Newborn and Child Health — Community engagement to improve awareness, and use of family planning products and services
  Other Names: Community Mobilization

SUMMARY:
Aim To evaluate the impact of an integrated Family Planning-Maternal,Newborn and Child Health service delivery model to increase coverage of MCM in a rural Pakistan.

Objectives

* To gain an understanding of the cultural and health service delivery contexts to inform a socio-culturally appropriate and acceptable intervention package scalable in rural Pakistan.
* To implement the intervention package at health facilities and outreach communities through existing public and private sector resources
* To measure the impact and level of effectiveness of interventions on the uptake MCM
* To identify and quantify the drivers of improved uptake of voluntary methods of FP especially MCM

DETAILED DESCRIPTION:
Interventions focusing on community outreach programs and interpersonal communications increase social acceptance of FP methods. However, home based counseling alone is not sufficient for the uptake and continuation of FP methods and developing linkages with health facilities and maintaining privacy at a health facility and being more culturally and religiously acceptable is also important. With this in mind, efforts have been made involving facility and community level health care providers for provision of MNCH services as the primary mandate of National Maternal Newborn and Child Health program. However, there are still deficiencies at inter and intra facility level, for example; a lack of coordination among departments such as Paediatrics and Gynecology & Obstetrics, lack of management level coordination with front line providers, lack of equipment and logistics management manifested as imbalance demand and supply and lack of overall governing bodies . Thus, overarching interventions covering service delivery platforms at facility and community levels necessitates the integration and scaling up of FP and MNCH services.

The theoretical underpinning of behavior change will be based on the Theoretical Domain Framework (TDF) v2.0. The TDF will be applied to provide an in-depth exploration and understanding of factors on the demand and supply side and their interaction with and influences on FP uptake. This project aims to implement a complex intervention (see figure 2) within health facilities and their catchment communities. This complex intervention includes a series of strategies involving community engagement by extensive community mobilization, availability of trained staff and sustainable supply of commodities with the required recording and reporting system. Continuous process monitoring and quality assurance will help to replicate the success and address possible barriers during implementation of the intervention. The mechanism of action built on the TDF adopts domains and constructs including, knowledge, skills, beliefs and intentions. Furthermore, the TDF provides a detailed understanding of complex behaviour thus will be used to evaluate the impact of complex interventions/ strategies.

Research Question What is the impact of integrating FP- MNCH services on uptake of voluntary modern contraceptive methods in a rural district of Sindh province, Pakistan?

ELIGIBILITY:
Inclusion Criteria:

* Healthy women of reproductive age living in the study areas

Exclusion Criteria:

* non resident living foe short term less than three months

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 125000 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
mCPR | 18 -24 Months
  Number of women age 15-49 years currently married who are using (or whose partner is using) a modern contraceptive method. (Modern methods include: male and female sterilization, injectable, intrauterine devices (IUDs), contraceptive pills, implants, male condoms, the standard days method, locational amenorrhea method, and emergency contraception)

SECONDARY OUTCOMES:
Unmet need | 18- 24 months
  Proportion of women who
  1. are not pregnant and not postpartum amenorrhea and are considered fecund and want to postpone their next birth for 2 or more years or stop childbearing altogether but are not using a contraceptive method, or
  2. have a mistimed or unwanted current pregnancy, or
  3. are postpartum amenorrhea and their last birth in the last 2 years was mistimed or unwanted.
Demand satisfied | 18- 24 months
  Proportion of demand satisfied by modern methods:
  Current contraceptive use (any modern method) divided by Unmet need + current contraceptive use (any method)
Women attitude towards family planning | 18- 24 months
  Proportion of women showing positive attitude towards FP
Unwanted pregnancy/births | 18- 24 months
  Planning status of births/pregnancies Women reported whether their births/pregnancies were wanted at the time (planned birth), at a later time (mistimed birth), or not at all (unwanted birth).
  Sample: Current pregnancies and births in the 5 years before the survey to women age 15-49
Inter-pregnancy Interval | 18- 24 months
  The number of months between a live birth and the conception of the next live birth. This was calculated by subtracting the "Date of last live birth" item from the date of birth to obtain a live-birth interval, then subtracting gestational age (months) of the birth from the live-birth interval.

CONTACTS AND LOCATIONS:
Locations (1):
- Aga Khan University, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Memon ZA, Reale S, Ahmed W, Spencer R, Lashari TH, Bhutta Z, Soltani H. Effects of Integrating Family Planning With Maternal, Newborn, and Child Health Services on Uptake of Voluntary Modern Contraceptive Methods in Rural Pakistan: Protocol for a Quasi-experimental Study. JMIR Res Protoc. 2022 Mar 8;11(3):e35291. doi: 10.2196/35291. PMID 35258461